CLINICAL TRIAL: NCT00335881
Title: Multicentre Study to Assess Persistence of Antibodies Against Hepatitis B & Immune Response to a Hepatitis B Challenge Dose in Healthy Children 4 to 6 Years Old Previously Vaccinated With 4 Doses of GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine
Brief Title: Persistence of the Immune Response to Hepatitis B in 4-6 Years Old Children Previously Vaccinated With DTPa-HBV-IPV/Hib
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106745
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
Keywords: Prophylaxis for hepatitis B disease
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: hepatitis B vaccine

SUMMARY:
Persistence of seroprotective antibody concentrations & immunological memory shown by the ability to mount a response to a challenge dose of HBV vaccine

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 4 to 6 years at the time of study entry .
* Subjects who have received a total of 4 doses of DTPa-HBV-IPV/Hib vaccine in previous vaccination studies.
* Evidence of previous hepatitis B booster vaccination or disease since administration of the fourth dose of DTPa-HBV-IPV/Hib vaccine.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2006-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentration

SECONDARY OUTCOMES:
Persistence of antibodies to the other DTPa-HBV-IPV/Hib vaccine antigens.
Sol & unsol symptoms after HBV vaccination, SAEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- Germany (31):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Freising, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Landsberg am Lech, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Schoeneberg - Kuebelberg, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Altenholz, Schleswig-Holstein
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Zinke M, Disselhoff J; DTP a-HBV-IPV-110 and -111 study groups; Gartner B, Jacquet JM. Immunological persistence in 4-6 and 7-9 year olds previously vaccinated in infancy with hexavalent DTPa-HBV-IPV/Hib. Hum Vaccin. 2010 Feb;6(2):189-93. doi: 10.4161/hv.6.2.10117. PMID 20009522
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register